CLINICAL TRIAL: NCT03279419
Title: Thermal Imaging of the Peripheral Vasculature in Liver Disease.
Brief Title: Thermal Imaging in Liver Disease.
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS ID 189169
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Liver disease: 15 patients with acute or chronic liver disease of any aetiology. Serial static images to be taken at up to 3 time points using thermal imaging camera. Video images using thermal camera will be used to capture warming of one hand after cooling.
  Patient may or may not be receiving terlipressin therapy.
  Interventions: Diagnostic Test: Thermal imaging
- Normal: 15 patients without liver disease, and without any other disease or drug known to affect the peripheral circulation.
  Serial static images to be taken at up to 3 time points using thermal imaging camera. Video images using thermal camera will be used to capture warming of one hand after cooling.
  Interventions: Diagnostic Test: Thermal imaging

INTERVENTIONS:
Diagnostic Test: Thermal imaging — Use of thermal imaging camera to capture images of peripheral vasculature (hands).

SUMMARY:
This is a feasibility study, to assess if thermal imaging and/or near infrared imaging will be useful in identifying changes in the peripheral circulation in patients with different stages of liver disease.

The aim of this study is to use new and advanced thermal imaging techniques to identify changes in the peripheral circulation and hand temperature in patients with liver disease. These changes could be used as a non-invasive marker of the severity and progression of liver disease. Thermal imaging will also be used to assess the changes in the peripheral vasculature with the use of terlipressin, a drug used as treatment for specific complications of liver disease.

Patients with acute or chronic liver disease from any aetiology will be recruited, along with patients without liver disease as healthy controls. Patients with disease or on drugs known to affect the peripheral vasculature will be excluded.

All studies will be performed in a ward setting in the Royal Infirmary of Edinburgh. The subjects will be required for up to three sessions, each lasting 30 minutes. The session will involve static thermal images being taken, and video images of the hands warming up after being cooled for 30 seconds in water at a temperature of 7 degrees Celsius. If the patient is receiving terlipressin therapy, static images will be taken before, during and after terlipressin therapy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic liver disease (any stage)
* diagnosis of acute liver disease (any aetiology)

Exclusion Criteria:

* on drugs known to affect peripheral circulation
* conditions known to affect peripheral circulation e.g. Raynauds

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-70 with acute or chronic liver disease
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in peripheral vasculature as assessed by thermal imaging | 2 years

SECONDARY OUTCOMES:
Changes in peripheral vasculature in response to terlipressin therapy. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Univerity of Edinburgh and NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No